CLINICAL TRIAL: NCT03188861
Title: Systematic Screening for Comorbid Psychological Conditions in Cardiac Ambulatory Care Sensitive Conditions (ACSC) Patients With Multimorbidity in the Emergency Departments (ED)
Brief Title: Systematic Screening for Comorbid Psychological Conditions in Cardiac ACSC Patients With Multimorbidity in the ED
Acronym: EMASPOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Martin Moeckel, Prof. Dr., Charite University, Berlin, Germany
Other Study IDs: EA1/363/16; 0133/17/ST3 (Other: Corporate Data Protection)
Record Dates: First submitted 2017-05-31; First posted 2017-06-16 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Depression; Anxiety; Somatoform Disorders; Alcohol Abuse
Keywords: mental health conditions in ACSC patients; multimorbidity; health care utilization
MeSH Terms: conditions — Depression; Anxiety Disorders; Somatoform Disorders; Alcoholism; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
EMASPOT assesses the prevalence and impact of mental health conditions in multimorbid emergency patients with cardiac ACSC on transsectoral utilisation of health care services.

DETAILED DESCRIPTION:
The specific aims of EMASPOT are primarily to determine the prevalence of mental health conditions (MHC) (i.e., symptoms of depression, anxiety, somatoform disorders, and alcohol abuse) in patients with multimorbidity and cardiac ACSC in a prospective cohort study.

The study population comprises patients admitted to an ED in Berlin-Mitte during the study period from 01.06.2017 to 31.05.2018 with cardiac complaints who are admitted to the hospital or discharged from ED. The study focusses especially on older and multimorbid patients. Multimorbidity is defined as the presence of more than two chronic diagnoses.

After having given informed consent patients are enrolled in the study and interviewed by a study nurse. Self-reported symptom burden for depression, anxiety disorders, somatoform disorders, alcohol abuse as well as frequency of utilization of health care services are assessed. Medical data will be abstracted from medical charts and include somatic comorbidities, medication and diagnostic procedures and interventions during hospitalization.

Individual semi-structured interviews will be conducted with 30 patients to assess the treatment expectations and underlying motives for ED-visits, as well as with 30 health care professionals to investigate perceptions of challenges regarding identification and treatment of patients with MHC.

All patients will have a 6-months follow-up after discharge from the ED. The follow-up is conducted either by telephone calls, e-mail or via mail. The follow-up data will include mental health conditions as assessed at baseline, frequency of utilization of health care services and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to one of the EDs in Berlin-Mitte due to cardiac complaints (acute heart failure, angina pectoris, dyspnea, arrhythmias)
* Age 50 and older

Exclusion Criteria:

* Age 49 and younger
* Inability to give written informed consent (cognitive impairment, legal guardianship)
* Insufficient language skills to complete the questionnaire in one of the provided languages (German, English, Russian, Turkish)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises patients admitted to an ED in Berlin-Mitte during the study period from 01.06.2017 to 31.05.2018 with cardiac complaints who are admitted to the hospital or discharged from ED. The study focusses especially on older and multimorbid patients. Multimorbidity is defined as the presence of more than two chronic diagnoses.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Mental health conditions | Baseline
  Proportion of patients with a high self-reported symptom burden for at least one of four mental conditions: depression, anxiety disorders, somatoform disorders, alcohol abuse

SECONDARY OUTCOMES:
Prevalence of mental disorders | Baseline
  Prevalence of mental disorders as assessed by structured clinical interview
Health outcomes | 6-months follow-up
  Patient-reported health outcomes after 6 months ((Mental health conditions: Depression, anxiety, somatoform symptoms, alcohol abuse) and Quality of life)
Utilization of health care systems | Baseline
  Frequency of health care system utilization before ED visit
Utilization of health care systems | 6-months follow-up
  Frequency of health care system utilization after ED visit
Expectations towards ED-care, semi-structured qualitative interviews | Baseline
  Patient (n≈30) and providers (n≈30) expectations towards ED-care and psychological care, assessed in a qualitative interview and categorized on the basis of qualitative methods

CONTACTS AND LOCATIONS:
Overall Officials: Martin Möckel, Prof. Dr., Principal Investigator — Division of Emergency Medicine, Charité University Hospital Berlin
Locations (1):
- Division of Emergency Medicine, Charité University Hospital, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schneider A, Wagenknecht A, Sydow H, Riedlinger D, Holzinger F, Figura A, Deutschbein J, Reinhold T, Pigorsch M, Stasun U, Schenk L, Mockel M. Primary and secondary data in emergency medicine health services research - a comparative analysis in a regional research network on multimorbid patients. BMC Med Res Methodol. 2023 Feb 4;23(1):34. doi: 10.1186/s12874-023-01855-2. PMID 36739382
- [Derived] Schneider A, Riedlinger D, Pigorsch M, Holzinger F, Deutschbein J, Keil T, Mockel M, Schenk L. Self-reported health and life satisfaction in older emergency department patients: sociodemographic, disease-related and care-specific associated factors. BMC Public Health. 2021 Jul 21;21(1):1440. doi: 10.1186/s12889-021-11439-8. PMID 34289829
- See also: project web page — http://emanet.charite.de